CLINICAL TRIAL: NCT02546219
Title: Investigating the Role of a4b7 Integrin as a Therapeutic Target in Eosinophilic Esophagitis
Brief Title: a4b7 Integrin in Eosinophilic Esophagitis
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John J. Garber III, MD, Assistant in Medicine, Massachusetts General Hospital
Other Study IDs: 2015P000816
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Eosinophilic Esophagitis
Keywords: eosinophilic esophagitis; EoE; integrins
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and esophageal eosinophils will be analyzed and may be stored for future studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with EoE: Adult patients with active eosinophilic esophagitis will under blood collection and esophagus biopsies in order to perform eosinophil isolation and characterization.
  Interventions: Other: Eosinophil isolation and characterization.

INTERVENTIONS:
Other: Eosinophil isolation and characterization. — Peripheral blood and esophageal biopsies will be obtained from study subjects for further analysis of eosinophils integrin profiles.

SUMMARY:
The overall objective of this preclinical study is to further the investigators mechanistic understanding of the role that the α4β7 and mucosal addressin cell adhesion molecule (MAdCAM-1) pathway plays in mediating eosinophil recruitment in EoE. To accomplish this, the investigators aim to (1) determine the baseline and dynamic patterns of α4β7 integrin expression on circulating and tissue eosinophils in EoE and in the setting of non-EoE esophageal eosinophilia (e.g., reflux esophagitis) and (2) determine the complete profile of eosinophil integrin molecules that may play a role in active EoE.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent
2. Male or female patients aged 18-65 years at time of screening
3. Confirmed active EoE at screening or within 8 weeks prior to baseline visit, as defined by esophageal mucosal eosinophils ≥15 per high power field (HPF, 400X magnification) despite at least 4 weeks of proton pump inhibitor (PPI) therapy with omeprazole 20 mg twice daily or the equivalent. updated 14APR2015 Page 8 of 19
4. Within the week prior to dosing, patient has one of the following symptoms of moderate, or worse, severity: dysphagia, vomiting, regurgitation, abdominal pain, chest pain/heartburn.
5. Maintained on a stabilized diet for at least 6 weeks prior to screening and during the course of the study; stable diet is defined as no initiation of single or multiple elimination diets or reintroduction of previously eliminated food groups.
6. Willing and able to comply with all clinic visits and study-related procedures
7. Able to understand and complete study-related questionnaires

Exclusion Criteria:

1. Another disorder that causes esophageal eosinophilia (e.g., hypereosinophilic syndrome, Churg-Strauss, parasitic infection)
2. History of abnormal gastric or duodenal biopsy or documented GI disorders other than EoE (e.g., celiac disease, Crohn's disease or H. pylori infection)
3. History of the following GI surgeries: fundoplication, gastric surgery or surgery for esophageal atresia
4. Use of systemic immunosuppressive or immunomodulating agents (oral prednisone, anti-immunoglobulin E (IgE) monoclonal antibody (mAb), methotrexate, cyclosporine, INFα, or anti-TNF) within six months prior to study entry.
5. A stricture on endoscopy that prevents passage of the endoscope
6. Participation in any investigational drug or device study within 30 days prior to study entry.
7. Female subjects who are pregnant or nursing.
8. Chronic infections such as HIV, hepatitis B or C, active mycobacterial (TB) or fungal infections.
9. Neoplasm or a history of malignancy in the preceding 5 years.
10. Concurrent infection or disease that may preclude assessment of eosinophilic esophagitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with active eosinophilic esophagitis
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of eosinophils expressing a4b7 integrin | 8 weeks
  Eosinophil expression levels of a4b7 integrin will be assessed on peripheral and esophageal eosinophils during active EoE and after treatment-induced remission.

CONTACTS AND LOCATIONS:
Overall Officials: John J Garber, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States